CLINICAL TRIAL: NCT03596112
Title: The Difference in Wound Size Reduction Comparing Two Frequently Used Wound Dressings in Everyday Care - a Randomized Controlled Trail
Brief Title: The Difference in Wound Size Reduction Comparing Two Frequently Used Wound Dressings in Everyday Care
Acronym: wound-size
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Responsible Party: Principal Investigator, Sebastian Probst, Prof Dr, School of Health Sciences Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Wound size reduction
Record Dates: First submitted 2018-07-10; First posted 2018-07-23 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-02

CONDITIONS: Wound Heal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- polyacrylate wound pad (Experimental): Use of cellulose and distinct layers of sodium-polyacrylate pad for wound care; frequency: twice a week
  Interventions: Other: application of a polyacrylate wound pad
- hydrocellular foam pad (Active Comparator): Use of standard foam pad for wound care; frequency: twice a week
  Interventions: Other: Hydrocellular foam

INTERVENTIONS:
Other: application of a polyacrylate wound pad — A sterile polyacrylate wound pad with activated carbon cloth treatment will be applied to chronic wounds in an outpatient clinic from a specialist nurse
  Arms: polyacrylate wound pad
Other: Hydrocellular foam — Active Comparator: hydrocellular foam pad serile hydrocellular standard foam pad will be applied to chronic wounds in an outpatient clinic from a specialist nurse
  Arms: hydrocellular foam pad

SUMMARY:
Chronic wounds (CW) such as leg or foot ulcers are slow healing wounds. They have a high recurrence rate and are associated with pain, infection, smell and exudate. The signs and symptoms of a chronic wounds are not only a burden on those who are affected by it but also on the health care system and society in general. With a prevalence of 1% in the general population, the prevalence rises to 3% in the over 80-age group. Current therapeutic approaches are multifaceted and focus on improving wound healing and preventing recurrences. Advanced wound dressings, especially super absorbent dressings are an important part of the wound care. Heavy wound exudate, if unabsorbed, may damage surrounding healthy skin and thus delay wound healing and contribute to maceration and excoriation regimen as CW may deliver excessive amounts of exudate followed by maldour. Maldodourous wounds can have a profoundly negative impact on the quality of life of the patient and of their carers causing feelings of guilt repulsion and leading to social isolation and depression. Therefore, it is important to use effective advanced wound dressings that are capable of managing wound exudate and with that promote wound healing. Currently the standard approches to managing exudate and wound odour are the use of hydrocellular foam dressing with silver or absorbent dressings like of a sterile polyacrylate wound pad with activated carbon cloth treatment. However, there is no evidence demonstrating whether there is adifference in wound size as an indicator of wound healing when comparing the application of a sterile polyacrylate wound pad with activated carbon clothtreatment to a standard non-adhesive hydrocellular foam dressing with silver treatment in a randomised controlled trail.

A randomized controlled trail with 90 participants in one wound care outpatient clinic is proposed.

Data will be analysed using SPSS version 23. Univariate and bivariate analysis will be conducted according to the data level and distribution.

This research project is designed to compare two wound dressings in everyday care. Since the cost of leg ulcers to individuals, the economy, and society is high, the evaluation of wound care dressings that leads to a reduction of wound size and promote wound healing are important for the individuals affected, their families, society at large and the health care system.

DETAILED DESCRIPTION:
Chronic wounds (CW) are poorly healing wounds (Persoon et al., 2004). Chronic leg (LU) and foot ulcers (DU) occur in many adults with vascular disease or diabetes and are attributed to chronic venous insufficiency, arterial disease, prolonged pressure, or neuropathy (Frykberg & Banks, 2015). Epidemiological data from industrialised countries including the United States of America and Scandinavian countries have shown that the prevalence of leg ulcers in the general population is 1%; while it is 3% in people over 80 years of age (Posnett, Gottrup, Lundgren, & Saal, 2009). If these findings are applied to the Swiss context then there are an estimated 80'000 to 90'000 VLU sufferers of which 8,000 persons are in the above-80 population segment (above 80 year population in Switzerland: 391,000 ) (Swiss Federal Statistical Office, 2016b). These ulcers last on average 12 to 13 months, recur in up to 60% to 70% of patients, can lead to loss of function and decreased quality of life, and are a significant cause of morbidity (Frykberg & Banks, 2015).

Predominantly a condition of the elderly, chronic wounds are becoming more prevalent and more difficult to treat and are associated with high treatment costs. The care for such conditions has been an estimated 2% to 3% of all health expenditures in developed countries (Posnett et al., 2009). With a Swiss health budget of 80 billion Swiss francs in 2016, this would translate into an annual cost up to 2.4 billion Swiss francs (Swiss Federal Statistical Office, 2016a).

.The care of chronic wounds has become its own specialty. The therapeutic approach to the management of CW is a multifaceted approach targeting the management of risk factors associated with healing rate and recurrence. Evidence showed the healing rate within a chronic wound is reported to be between 0.1 cm2 and 1cm2 per week independent of the wound-type (Hussain, 2015). The healing rate is mostly associated of the management of bacteria that is amongst other things manifested in wound odour and the used wound dressing and its absorption of wound exudate(Probst, 2015).

Wound odour is not attributed to any one particular source but is thought to be caused by a combination of bacteria including aerobic and anaerobic species, necrotic tissue, poorly vascularized tissue and light levels of exudate (Gethin, Grocott, Probst, & Clarke, 2014). Malodour due to wounds can have a profoundly negative impact on the quality of life of the patient and of their carers causing feelings of guilt repulsion and leading to social isolation and depression (Gethin et al., 2014).

Wound exudate is a normal part of the wound healing process in any kind of wound. In general, the quantity of exudate produced decreases as the wound heals and progresses towards wound closure (Probst & Huljev, 2013). Exudate is particularly noticeable during the inflammatory and proliferative phases of healing because it provides nutrients as an energy source for metabolizing cells and plays a role in regulating the moisture level in the local wound environment (Coleridge-Smith, Lok, & Ramelet, 2005). This is the case in all chronic wounds. Managing a wound with a high level of exudate is one of the most commonly cited clinical problems not only in LU but also in DU or pressure ulcers (Chamanga, 2015; Probst, 2015; Tickle, 2015). High levels of exudate are challenging in terms of the selection of wound dressing products capable of handling the fluid levels and also the prevention of damage to the surrounding healthy skin (Tickle, 2015). Leakage of exudate through the dressing not only increases the risk of maceration or/ and cross-infection, it may also be distressing for the patient because of soiling of clothing and bedding and possible malodor (Probst, Arber, & Faithfull, 2013b).Due to unabsorbed heavy exudate, healing is delayed and surrounding skin can be badly damaged due to maceration and excoriation (Chamanga, 2015). Additionally, the psychological effects of coping with a chronic wound on a day to day basis should not be underestimated (Probst, Arber, & Faithfull, 2013a). For health services, the management of excess exudate presents considerable costs in terms of health professionals' time spent on more frequent visits to change dressings and costs for dressings and associated preventive measures such as skin protection (Probst, 2015). Therefore, the use of effective advanced wound dressings that manage exudate are an important aspect of wound therapy. There are many advanced wound dressings on the market absorbing excessive amounts of exudate. Currently the standard approaches to managing exudate and the presence of high bacteria load are dressings with silver such as the use of hydrocellular foam dressing with silver (non-adhesive or adhesive) or absorbent dressings. However, there is no evidence demonstrating the difference of wound size applying a sterile polyacrylate wound pad with activated carbon cloth treatment in comparison to a standard non -adhesive hydrocellular foam dressing with silver treatment.

This research project is designed to compare two wound dressings in everyday care. Through this comparison the effective amount of wound exudate in the population of LU and DU can be measured. Since the cost of leg ulcers to individuals, the economy, and society is high, the evaluation of wound care dressings that leads to a reduction of wound size and promote wound healing are important for the individuals affected, for society at large and the health care system.

ELIGIBILITY:
Inclusion Criteria:

* existing leg ulcer or diabetic foot ulcer
* Light to heavy exudating wounds
* Age over 18 years
* Proficiency in the French language

Exclusion Criteria:

* Valid informed consent is not or cannot be given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
change of wound size | 12 weeks
  the wound-size (in cm2) of the target ulcers will differ by 20% over a 12 weeks treatment period between patients with LU and DU using a sterile polyacrylate wound pad with activated carbon cloth treatment and a standard non-adhesive hydrocellular foam dressing with silver treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian E Probst, Prof Dr, Principal Investigator — University of Applied Sciences and Arts Western Switzerland
Locations (1):
- Cité Génération Maison de santé, Onex, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No
data will be anonymised